CLINICAL TRIAL: NCT03108183
Title: A Prospective Study to Evaluate the Longterm Treatment Results After Micro-surgical Root Resection of Teeth With Post and Core and Crown
Brief Title: Apicoectomy Longterm Results
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Angel; 29-214 ex 16/17 (Other: Ethics committee Medical University of Graz)
Record Dates: First submitted 2017-03-17; First posted 2017-04-11 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Periapical Diseases
MeSH Terms: conditions — Periapical Diseases | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: x-rays — To get further and actual information about periapical lesions, different x-rays will be done (panoramic radiographic, small picture ray, cone beam computed tomography). Furthermore a periodontal status will be performed.

SUMMARY:
The purpose of the study is to evaluate the longterm treatment results after micro-surgical root resection of teeth with post and core and crown.

DETAILED DESCRIPTION:
All 73 patients, who have been treated with apicoectomy on teeth with post and core and crown between the years 2004 and 2006 and who have already been followed up in 2008, will be followed up once more in 2017.

The patients will have a clinical and radiologic examination. The investigators will examine if new periapical lesions, bone loss, fracture of teeth or loss of teeth exist.

ELIGIBILITY:
Inclusion Criteria:

* All 73 patients, who were treated with apicoectomy on teeth with post and core and crown between the years 2004 and 2006 and who have already been followed up in 2008, will be followed up once more in 2017.

Exclusion Criteria:

* Pregnancy
* Patients who do not want to participate in clinical and radiological follow up.

Ages: 27 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 73 patients, who have been treated with apicoectomy on teeth with post and core and crown between the years 2004 and 2006 and who have already been followed up in 2008, will be followed up once more in 2017.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Appearance of periapical lesions on tooth after root resection | 1 day
  Appearance assessed by X-ray and classified according to Molven et al. (1987)
Size of periapical lesions on tooth after root resection | 1 day
  Size assessed by X-ray and classified according to Molven et al. (1987)

SECONDARY OUTCOMES:
Vertical and horizontal bone loss on the tooth after root resection | 1 day
  Bone loss in mm assessed by X-ray and probing
Occurrence of tooth fractures | 1 day
  Number of tooth fractures assessed by X-ray
Occurrence of tooth loss | 1 day
  Number of tooth losses assessed by clinical and radiological evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Jakse, MD, Principal Investigator — Department of dental medicine and oral health, Medical University of Graz
Locations (1):
- Medical University, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molven O, Halse A, Grung B. Observer strategy and the radiographic classification of healing after endodontic surgery. Int J Oral Maxillofac Surg. 1987 Aug;16(4):432-9. doi: 10.1016/s0901-5027(87)80080-2. PMID 3117915